CLINICAL TRIAL: NCT02993341
Title: Topical Tranexamic Acid (TXA) in Hip Fractures, A Double-Blind, Randomized Controlled Trial
Brief Title: Topical Tranexamic Acid (TXA) in Hip Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sault Area Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TXA-WASH-01
Record Dates: First submitted 2016-04-12; First posted 2016-12-15 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hip Fracture; Anemia
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid Wash (Experimental): Participants in the experimental arm will receive a wash of tranexamic acid topically at the site of surgery.
  Interventions: Drug: Tranexamic Acid
- Saline Wash (Placebo Comparator): Participants in the control arm will receive a wash of saline topically at the site of surgery.
  Interventions: Other: Saline Wash

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid Wash
Other: Saline Wash
  Arms: Saline Wash

SUMMARY:
Mechanisms by which to reduce exposure to allogeneic blood are of financial and clinical benefit in the hip fracture population. Tranexamic acid (TXA) is an inexpensive medication with low complication risk. Its use in the hip fracture population is unproven. The purpose of this study is to evaluate the efficacy and safety of topical tranexamic acid in reduction of peri-operative blood loss in hip fracture surgery.

DETAILED DESCRIPTION:
The results of this study may dramatically alter the manner in which surgeons manage hip fracture patients in Canada. The use of topical TXA in operatively-treated hip fracture patients has the potential to reduce perioperative blood loss and consequently reduce exposure to allogeneic blood transfusion. This will positively influence post-operative morbidity and mortality, while at the same time substantially reduce hospital length of stay and overall health care costs. The proposed study is felt to have minimal risk, and is a relatively inexpensive study.

Update: An interim analysis was completed in January 2018. The Data Safety Monitoring Committee reviewed the results and recommend the trial continue as planned.

The final data analysis is in process. The abstract will be uploaded upon completion.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met to be eligible:

1. 18 years of age or older
2. Diagnosis of hip fracture (Intracapsular, Intratrochanteric or Subtrochanteric) requiring surgical repair
3. Patient/surrogate decision maker provide signed informed consent

Exclusion Criteria:

Participants cannot be included in this study if any of the following criteria apply:

1. Patient has documented renal failure with glomerular filtration rate of <30ml/min/1.73m2
2. Documented allergy to tranexamic acid
3. Current use of hormone replacement therapy
4. Acquired disturbances of colour vision
5. Refusal of blood products
6. Pre-operative use of anticoagulant therapy (Coumadin, heparin < 5 days of surgery, fibrinolytic disorders requiring intraoperative anti-fibrinolytic treatment)
7. Coagulopathy (pre-operative platelet count <150,000/mm3, International Normalized Ratio (INR) >1.4, prolonged Partial Thromboplastin Time (PTT) >1.4x normal)
8. Hematuria
9. Acute coronary syndrome within 6 weeks of fracture
10. Any history of venous thromboembolism
11. Any intraoperative surgical/medical/anesthetic complications i.e.: myocardial infarction or neurovascular injury occurring prior to application of the tranexamic acid
12. Pregnant or lactating
13. Any major medical or psychiatric disorder that in the opinion of the investigator, might prevent the subject from completely participating in the study or interfere with the interpretation of the study results
14. Unable/unwilling to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-11; Primary Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | 1 day and 3 days post-surgery
  change in hemoglobin levels day 1 and 3 post-op compared to pre-op values and need for allogenic blood transfusion up to 3 days post-op

SECONDARY OUTCOMES:
All-cause mortality | 30 days post-surgery
Reduced risk of thrombotic event | 30 days post-surgery
  Measure incidence of venous thromboembolism (symptomatic ultrasound proven deep vein thrombosis or pulmonary embolism diagnosed by a ventilation-perfusion scan or computed tomography angiogram)
Reduced peri-operative complications | 30 days post-surgery
  (post-operative surgical site infection, acute coronary syndrome, cerebrovascular event)

CONTACTS AND LOCATIONS:
Locations (1):
- Sault Area Hospital, Sault Ste. Marie, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costain D, Elder G, Fraser B, Slagel B, Kelly A, Cheong Y, Fera L. Topical tranexamic acid in hip fractures: a randomized, placebo-controlled double-blinded study. Can J Surg. 2021 Aug 10;64(4):E449-E456. doi: 10.1503/cjs.014220. Epub 2021 Aug 1. PMID 34388107